CLINICAL TRIAL: NCT07338539
Title: BIOlogically-guided Short-course HypOfractionatedRadiation Therapy in Poor-prognosis GBM (BIO-SHORT): A Prospective Phase 2 Randomised Control Trial
Brief Title: BIO-SHORT: Biologically Guided Short-Course Hypofractionated RT for Poor-Prognosis GBM
Acronym: BIO-SHORT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4840
Record Dates: First submitted 2025-11-24; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, open-label2-arm Phase 2 randomized controlled trial with a superiority design. The standard arm will comprise of 3 week hypo-fractionated RT(40Gy/15#).The test arms will comprise of dose escalated hypo-fractionated RT (5 fractions/10 fractions). The usage of TMZ will be standard across both arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Arm (Active Comparator): The standard arm will comprise of 3 week hypo-fractionated RT(40Gy/15#).
  Interventions: Radiation: Standard radiotherapy using hypofractionated RT
- Dose-escalated hypofractionated RT (Experimental): Patients in the experimental arm will undergo pretreatment evaluation, MRI-based simulation, and radiotherapy delivery similar to the standard arm, with the addition of pre-treatment F-DOPA PET imaging performed according to institutional consensus protocols. Biological target volumes (BTVs) will be delineated using a tumor-to-white-matter uptake ratio >2.0.
  The initial clinical target volume (CTV-initial) will include the BTV, postoperative cavity, contrast-enhancing tumor on T1-weighted MRI, and gross disease. A 1.5-cm margin, edited for anatomical barriers, will generate the CTV-final to account for infiltrative spread. The planning target volume (PTV) will be created using a 3-5-mm geometric expansion.
  Dose prescription will be based on PTV volume and location. Patients with PTV >30 cc or tumors not involving the brainstem will receive 40 Gy in 10 fractions to the BTV and 35 Gy in 10 fractions to the PTV. Those with PTV ≤30 cc or brainstem involvement will receive 30 Gy in 5 fra
  Interventions: Radiation: Experimental Arm Intervention

INTERVENTIONS:
Radiation: Standard radiotherapy using hypofractionated RT — Patients in the standard arm will undergo target volume delineation using conventional imaging. The initial clinical target volume (CTV-initial) will include the postoperative cavity, contrast-enhancing tumor on T1-weighted MRI, and gross disease. A 1-cm isotropic expansion, edited for anatomical barriers, will generate the CTV-final to account for infiltrative spread. The planning target volume (PTV) will be created using a 3-mm geometric margin for setup uncertainty. Radiotherapy will be delivered using photon-based image-guided IMRT, prescribed to a total dose of 40 Gy in 15 fractions, administered five days per week.
  Arms: Standard Arm
Radiation: Experimental Arm Intervention — Patients in the experimental arm will undergo pretreatment evaluation, MRI-based simulation, and radiotherapy delivery similar to the standard arm, with the addition of pre-treatment F-DOPA PET imaging performed according to institutional consensus protocols. Biological target volumes (BTVs) will be delineated using a tumor-to-white-matter uptake ratio >2.0.
  The initial clinical target volume (CTV-initial) will include the BTV, postoperative cavity, contrast-enhancing tumor on T1-weighted MRI, and gross disease. A 1.5-cm margin, edited for anatomical barriers, will generate the CTV-final to account for infiltrative spread. The planning target volume (PTV) will be created using a 3-5-mm geometric expansion.
  Dose prescription will be based on PTV volume and location. Patients with PTV >30 cc or tumors not involving the brainstem will receive 40 Gy in 10 fractions to the BTV and 35 Gy in 10 fractions to the PTV. Those with PTV ≤30 cc or brainstem involvement will receive 30 Gy in 5 frac
  Arms: Dose-escalated hypofractionated RT

SUMMARY:
High grade gliomas, particularly glioblastoma, are among the most aggressive brain tumors and are associated with poor outcomes despite standard treatment. Many patients, especially older adults or those with poor general health, are not suitable for surgery and have a life expectancy of less than 12 months. Current standard includes a shortened course of radiotherapy (over 3 weeks) combined with chemotherapy using temozolomide (TMZ), which offers limited survival benefits. This study aims to explore whether delivering radiotherapy in a shorter duration (1 or 2 weeks) at a higher dose, guided by advanced imaging with a PET scan, can improve survival in this group of patients. PET scans help identify the most active parts of the tumor, which aids in targeting of these areas more precisely, potentially improving outcomes while reducing harm to healthy brain tissue. This study will randomly assign 116 eligible patients into two groups:

* One group will receive the current standard of care (3-week radiotherapy + TMZ).
* The other group will receive PET-guided radiotherapy over a shorter duration (either 5 or 10 sessions) at a higher dose, alongside TMZ.

The primary goal is to compare overall survival at one year between the two groups. The study will also assess how the disease progresses, side effects of treatment, and the impact on patients' quality of life. The study will be conducted over a total period of 6 years, including 4 years for patient enrolment and 2 years of follow-up. Participation in the study is entirely voluntary, and all patients will undergo an informed consent process. The study has been designed to follow all applicable ethical and regulatory guidelines. The results may help establish a more effective and convenient treatment option for patients with aggressive brain tumors and poor prognosis.

DETAILED DESCRIPTION:
Introduction:

Glioblastoma Multiforme(GBM) is the most common malignant primary brain tumor which is uniformly fatal with dismal long term survival rates despite aggressive multimodality therapy. A large proportion of the patients are elderly, presenting at over 65 years of age and their treatment is associated with even more inferior outcomes. Treatment of such elderly patients with typical normo-fractionated Radiotherapy (RT) {1.8-2Gy per fractionation} over 6-6.5 weeks leads to unnecessary protraction of treatment, unduly encumbering patients and their caregivers. Randomised trials and subsequent meta-analyses have shown that hypo-fractionated RT ( typically delivered over 2 -3 weeks ) achieves similar survival as longer 6 week schedules in elderly patients in poor general condition. Addition of Temozolomide based chemotherapy was subsequently shown to improve survival and in current practice hypo-ractionated short course RT(hypo-RT) with TMZ represents the most optimal management of GBM in the elderly achieving a median survival in the vicinity of 6-9 months. Similar survival has been reported in institutional series in poor prognosis High Grade Glioma. Cumulatively, all the data serve as a relatively homogenous point for providing benchmark outcomes which may be used to improve survival by means of treatment intensification and optimisation of the HypoRT -TMZ backbone in this setting.

One of the most tangible ways in which outcomes can be improved pertains to the usage of a higher cumulative RT dose. Retrospective institutional data suggest that normo-fractionated schedules (59.4Gy/33#) delivered in fit elderly individuals are associated with survival benefit. Concurrent data shows that similar increase in median survival to 14-15 months is achievable by the usage of 3 week hypofractionated regimens which are iso-effective to the Stupp regimen. Further safe reduction to a 2 week schedule has been shown in a recent trial using proton therapy and Positron Emission Tomography (PET) guided sub-volume dose escalation. The reduction of dose to the normal brain has shown to be more pragmatically achievable in a recent trial incorporating reduced margins (5mm as opposed to 1.5 -2 cm) for microscopic disease and photon based fractionated radiosurgery which achieved a median survival of 14.8 months with no compromised survival due to marginal recurrences. Overall there is a need for a pragmatic trial incorporating an abbreviated schedule of photon based hypo-fractionated RT (5 fractions/10 fractions) in poor prognosis High Grade Glioma (HGG) using reduced margins and PET based biological sub-volume boosting to deliver adequate doses to the gross tumor and minimise surrounding normal brain RT doses to improve median benchmark survival to 14-15 months as compared to the prevailing standard of care (40Gy/15# with temozolomide). The current trial plans to address this knowledge gap.

Primary Endpoint:

The primary endpoint will be the Overall Survival (OS) at 1 year. Overall Survival will be defined as the time elapsed from the date of randomization to date of death due to any cause.

Secondary Endpoint:

* Progression Free Survival (PFS) at 1 year- Progression Free Survival will be defined as the time elapsed from the date of randomization to the date of clinico-radiological progression or death.
* Toxicity assessment with the NCI Common Terminology Criteria for Adverse Events version 5 (CTCAE v5)
* Quality of life indices using the EORTC QLQC- 30 and its BN -20 module
* Quality of life without symptoms or toxicity in three health states TOX (toxicity), TWIST (time without symptoms) and REL (relapse)

Study Design:

The study will be a prospective, open-label2-arm Phase 2 randomized controlled trial with a superiority design. The standard arm will comprise of 3 week hypo-fractionated RT(40Gy/15#).The test arms will comprise of dose escalated hypo-fractionated RT (5 fractions/10 fractions). The usage of TMZ will be standard across both arms.

Study setting: The study will be conducted in the department of Radiation Oncology, Neuro Oncology Disease management group

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven IDH- wild type GBM or imaging defined GBM
* Neurological Predictor Scale (NPS) = 2-3
* Unfit for surgery and referred for direct RT
* Age >/= 50 years

Exclusion Criteria:

* IDH mutant glioma
* Histone altered glioma
* Multifocal disease or Gliomatosis like appearance which necessitates whole brain RT
* Disseminated disease in brain or spine
* NPS = 0-1 or = 4
* Karnofsky Performance Status score less than 50(Patient requires considerable assistance and frequent medical care)
* Prior administration of any systemic therapy directed against glioma (eg.Temozolomide, CCNU, Bevacizumab)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2031-10-27 (Estimated); Study Completion 2031-10-27 (Estimated)

PRIMARY OUTCOMES:
Survival Outcomes | 1 year
  . Overall Survival will be defined as the time elapsed from the date of randomization to date of death due to any cause.

SECONDARY OUTCOMES:
Survival Outcome | 1 year
  Progression Free Survival (PFS) will be defined as the time elapsed fromthe date of randomization to the date of clinico-radiological progression or death.
Quality of life indices | Baseline / Pre-radiotherapy, 4-6 weeks post-radiotherapy, 1 month, 3 months, 6 months, 9 months, and 12 months post-radiotherapy
  Quality of life indices using the EORTC QLQC- 30 and its BN -20 module
QTWiST (Quality of life Without Symptoms or Toxicity) calculation | will be done at 3 months
  Quality of life without symptoms or toxicity in three health states TOX (toxicity), TWIST (time without symptoms) and REL (relapse)
Toxicity Assessment | Baseline / Pre-radiotherapy, 4-6 weeks post-radiotherapy, 1 month, 3 months, 6 months, 9 months, and 12 months post-radiotherapy
  Toxicity assessment with the NCI Common Terminology Criteria for Adverse Events version 5 (CTCAE v5)- Grade 1-5

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No